CLINICAL TRIAL: NCT02965014
Title: Young Women-Focused HIV Prevention: Seek & Test in North Carolina (NC) Clinics
Brief Title: NC Young Women's CoOp
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the COVID-19 pandemic, this health department-based trial ended early to limit utilizing clinic services and resources and to ensure participant and staff safety. This termination primarily affected the 12-month follow-up appointments.
Sponsor: RTI International (Other)
Collaborators: Durham County Department of Public Health (Unknown); Guilford County Department of Public Health (Unknown); Wake County Human Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: R01DA041009 (NIH)
Record Dates: First submitted 2016-11-14; First posted 2016-11-16 (Estimated); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Condomless Sex; Human Immunodeficiency Virus (HIV); Sexually Transmitted Infection (STI); Alcohol and Drug Use
Keywords: Human Immunodeficiency Virus (HIV); Sexually transmitted infections (STI); mHealth; Substance abuse; Violence; Victimization; Sexual Risk
MeSH Terms: conditions — Unsafe Sex; Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Face-to-Face Young Women's CoOp (YWC) (Experimental): Participants in this arm will be offered a two-session face-to-face Young Women's CoOp (YWC) intervention.
  Interventions: Behavioral: Face-to-Face Young Women's CoOp (YWC)
- mHealth Young Women's CoOp (YWC) (Experimental): Participants in this arm will be offered training on the mobile health application mHealth Young Women's CoOp (YWC) and offered tablets with the mHealth application to complete the two-session intervention.
  Interventions: Behavioral: mHealth Young Women's CoOp (YWC)
- HIV Counseling and Testing (Active Comparator): Participants will be offered standard HIV counseling and testing services.
  Interventions: Behavioral: HIV Counseling and Testing

INTERVENTIONS:
Behavioral: Face-to-Face Young Women's CoOp (YWC) — Participants will be offered HIV counseling and testing (HCT) and a two-session face-to-face YWC intervention. The face-to-face sessions will include information addressing the intersection of substance use, sexual risk, and violence through skill building, role-play, and rehearsal.
  Arms: Face-to-Face Young Women's CoOp (YWC)
Behavioral: mHealth Young Women's CoOp (YWC) — Participants will be offered HIV counseling and testing (HCT) and training on the mHealth application, which will include all content addressed in the face-to-face YWC delivery format. Participants will also be offered a tablet to complete the two-session intervention.
  Arms: mHealth Young Women's CoOp (YWC)
Behavioral: HIV Counseling and Testing — Participants will be offered standard HIV counseling and testing (HCT).
  Arms: HIV Counseling and Testing

SUMMARY:
This three-arm cross-over randomized trial will develop, test, and compare the efficacy of two delivery formats of the Young Women's CoOp (YWC), which is designed to provide risk reduction and empowerment skills, as well as linkages to healthcare services for women who use substances. The current study will develop a revised version of the YWC and evaluate the relative efficacy of a face-to-face (face-to-face YWC), mobile Health application (mHealth YWC) delivery format, and HIV counseling and testing (HCT) as a control to reduce risky sexual behaviors and reduce substance use among young (18-25) African American women who use substances and are sexually active and have not recently been tested for HIV in three NC counties.

DETAILED DESCRIPTION:
The purpose of this study is to use the seek, test, treat, and retain framework to develop and test the efficacy of a clinic-based, age-appropriate, woman-focused HIV risk-reduction intervention to reduce sexual risk among up to 700 young sexually active African American women aged 18 to 25 who use drugs in three North Carolina counties. The researchers will test the delivery of the woman-focused intervention conducted in two formats, face-to-face YWC and mHealth YWC, using a three-arm cross-over randomized design in which counties are randomized to (1) HCT as the control, (2) face-to-face YWC; and (3) mHealth YWC that will be delivered on tablets using an interactive app. The researchers will fulfill the purpose of this study through the following aims: (Aim 1) To develop a new YWC intervention and recruitment strategies using formative methods to engage young African American women who use substances and have not recently been tested for HIV, clinic staff, and stakeholders to ensure age appropriateness, to identify barriers to reaching these young women and the challenges in conducting the intervention in the clinics, and to develop the mHealth YWC; (Aim 2) To test the efficacy of two formats of the woman-focused intervention program (face-to-face YWC and mHealth YWC) relative to HCT with up to 700 young women aged 18 to 25 in three North Carolina county health departments for primary outcomes at 6-, and 12-month follow-up assessments; (Aim 3) To estimate the total costs of implementing the face-to-face YWC and mHealth YWC interventions, and to assess the resource components that drive these costs; and (Aim 4) To examine the extent to which the face-to-face YWC and mHealth YWC are perceived by collaborating health clinic staff and participants as being acceptable and sustainable.

ELIGIBILITY:
Selected Inclusion Criteria:

* Identify as female
* Identify as Black or African American
* 18-25 years of age
* Have used alcohol or drugs in greater quantity or for a longer period of time than intended within the past 30 days

Exclusion Criteria:

* Participants may not be non-Black/African American

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 652 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Condomless Sex | Baseline
  Self-reported frequency of condomless sex
Condomless Sex | 6-month follow-up
  Self-reported frequency of condomless sex
Condomless Sex | 12-month follow-up
  Self-reported frequency of condomless sex
Frequency of Substance Use | Baseline
  Frequency of using illicit drugs and alcohol
Frequency of Substance Use | 6-month follow-up
  Frequency of using illicit drugs and alcohol
Frequency of Substance Use | 12-month follow-up
  Frequency of using illicit drugs and alcohol

SECONDARY OUTCOMES:
Increased Sexual Negotiation | Baseline
  Self-reported ability to negotiate condom use and other safe sexual behavior with a male partner
Increased Sexual Negotiation | 6-month follow-up
  Self-reported ability to negotiate condom use and other safe sexual behavior with a male partner
Increased Sexual Negotiation | 12-month follow-up
  Self-reported ability to negotiate condom use and other safe sexual behavior with a male partner
Reduced Alcohol and Illicit Drug Use for a Subsample of Participants | Baseline
  Self-reported amount of alcohol consumption and drugs used; Urine drug screen will be used to test for recent illicit drug use; Breathalyzer test results will be used to assess recent alcohol use
Reduced Alcohol and Illicit Drug Use for a Subsample of Participants | 6-month follow-up
  Self-reported amount of alcohol consumption and drugs used; Urine drug screen will be used to test for recent illicit drug use; Breathalyzer test results will be used to assess recent alcohol use
Reduced Alcohol and Illicit Drug Use for a Subsample of Participants | 12-month follow-up
  Self-reported amount of alcohol consumption and drugs used; Urine drug screen will be used to test for recent illicit drug use; Breathalyzer test results will be used to assess recent alcohol use
Reduced Violence and Victimization for a Subsample of Participants | Baseline
  Self-reported experiences of emotional, physical, and sexual abuse
Reduced Violence and Victimization for a Subsample of Participants | 6-month follow-up
  Self-reported experiences of emotional, physical, and sexual abuse
Reduced Violence and Victimization for a Subsample of Participants | 12-month follow-up
  Self-reported experiences of emotional, physical, and sexual abuse

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Browne, ScD, Principal Investigator — RTI International
Locations (4):
- United States (4):
  - Durham County Department of Public Health, Durham, North Carolina
  - Guilford County Department of Public Health - Greensboro, Greensboro, North Carolina
  - Guilford County Department of Public Health - High Point, High Point, North Carolina
  - Wake County Human Services, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Analytic data sets will be prepared in accordance with the "Privacy Rule" of the Health Insurance Portability and Accountability Act (HIPAA; http://www.hhs.gov/ocr/) as "limited data sets" in which names and other personal health identifiers are removed, birthdays have been converted to age at intake, and other dates have been changed to be days before or after the date of intake. Because there are fewer than 20,000 people in the data set, HIPAA says we cannot ensure that it is completely "de-identified"; consequently, HIPAA requires that we treat it as a "limited data set" and that we have a data sharing agreement (DSA) in place before giving anyone access to the client-level data. After the main findings are published, we will welcome other researchers who want to analyze the data in other ways. Requesting access to data will involve drafting an abstract, checking the feasibility relative to the available data, and seeking the permission of the PI and her team.

REFERENCES:
- [Result] Browne FA, Washio Y, Zule WA, Wechsberg WM. HIV-related risk among justice-involved young African American women in the U.S. South. Health Justice. 2023 Aug 24;11(1):32. doi: 10.1186/s40352-023-00228-7. PMID 37615878
- [Result] Osakwe CE, van der Drift I, Opper CA, Zule WA, Browne FA, Wechsberg WM. Condom Use at Last Sex and Sexual Negotiation Among Young African American Women in North Carolina: Context or Personal Agency. J Racial Ethn Health Disparities. 2024 Aug;11(4):2256-2264. doi: 10.1007/s40615-023-01693-4. Epub 2023 Jul 26. PMID 37495904
- [Result] Watkins RL, Browne FA, Kizakevich PN, Howard BN, Turner LB, Eckhoff R, Wechsberg WM. An Evidence-Based HIV Risk-Reduction Intervention for Young African American Women in the US South Using mHealth: Adaptation and Development Study. JMIR Form Res. 2022 May 9;6(5):e34041. doi: 10.2196/34041. PMID 35532978
- [Derived] Opper CA, Browne FA, Howard BN, Zule WA, Wechsberg WM. Assessing Differences in mHealth Usability and App Experiences Among Young African American Women: Secondary Analysis of a Randomized Controlled Trial. JMIR Hum Factors. 2024 Apr 16;11:e51518. doi: 10.2196/51518. PMID 38625721
- [Derived] Browne FA, Wechsberg WM, Kizakevich PN, Zule WA, Bonner CP, Madison AN, Howard BN, Turner LB. mHealth versus face-to-face: study protocol for a randomized trial to test a gender-focused intervention for young African American women at risk for HIV in North Carolina. BMC Public Health. 2018 Aug 6;18(1):982. doi: 10.1186/s12889-018-5796-8. PMID 30081868